CLINICAL TRIAL: NCT00895869
Title: Pain in Neonates During Screening for Retinopathy of Prematurity Using Binocular Indirect Ophthalmoscopy and Wide-field Digital Retinal Imaging: a Randomized Comparison
Brief Title: Pain in Neonates During Screening for Retinopathy of Prematurity Using Two Methods
Acronym: RETCAM
Status: Completed | Type: Observational
Sponsor: NHS Lothian (Other Government)
Responsible Party: Sponsor
Other Study IDs: BF01; JB001; RF001
Record Dates: First submitted 2009-05-07; First posted 2009-05-08 (Estimated); Last update posted 2024-09-23 (Actual); Status verified 2010-02

CONDITIONS: Retinopathy of Prematurity; Pain
Keywords: Screening; Retinopathy; Prematurity; Pain
MeSH Terms: conditions — Retinopathy of Prematurity; Pain; Retinal Diseases; Premature Birth

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Retinopathy of prematurity screening is painful. Wide field digital retinal imaging (WFDRI) and binocular indirect ophthalmoscopy (BIO) are being used for screening examinations. The aim of Edinburgh, UK based study is to compare the pain experienced by infants using both examination techniques.

DETAILED DESCRIPTION:
Infants undergoing routine eye screening at Edinburgh Royal Infirmary Neonatal Intensive Care Unit are to be recruited. Infants will be excluded if they require mechanical ventilation or analgesic medication or if they have moderate/severe neurological impairment. The first screening examination for each baby was included. Infants' eyes will be examined by both WFDRI and BIO with eyelid speculum by 2 experienced pediatric ophthalmologists in random order. Observations will be video-recorded during examinations to generate a pain score (premature infant pain profile) for both WFDRI and BIO. The pain scores, heart rates, oxygen saturations and time taken for WFDRI and BIO will be compared using paired t tests.

ELIGIBILITY:
Inclusion Criteria:

* Infants born at less than 32 weeks gestation and/or birth weight of less than 1500g.

Exclusion Criteria:

* Infants requiring mechanical ventilation
* Infants requiring analgesic medication
* Infants with moderate/sever neurological impairment

Max Age: 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Premature infants
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2004-04; Primary Completion 2008-01 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr B Fleck, MBChB FRCOpth BSc(Hons) MD, Study Chair — NHS Lothian; Dr C Dhaliwal, BSc(Hons) MBChB MRCPCH, Principal Investigator — NHS Lothian
Locations (1):
- NHS Lothian, Edinburgh, United Kingdom